CLINICAL TRIAL: NCT05077826
Title: Modern Energetic Methods of Response Improvement (MEMORI)
Brief Title: Enhancing Memory in Mild Cognitive Impairment and Early Stage Alzheimer's Disease
Acronym: MEMORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-203
Record Dates: First submitted 2021-09-07; First posted 2021-10-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Dementia; Memory; Transcranial direct current stimulation (tDCS); Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Full Current tES (Experimental): TES delivered with the anode over the right temple and cathode on the left arm, at an intensity of up to 4 milliamps, delivered for up to 40 minutes.
  Interventions: Device: North Coast Medical Activadose II
- Partial Current tES (Placebo Comparator): TES delivered with the anode over the right temple and cathode on the left arm, at an intensity of 0.1 milliamp, delivered for up to 40 minutes.
  Interventions: Device: North Coast Medical Activadose II

INTERVENTIONS:
Device: North Coast Medical Activadose II — tES device model Activadose II (North Coast Medical, Morgan Hill, CA, USA) programed to deliver tES.

SUMMARY:
The investigators have developed a low-risk transcranial Electrical Stimulation (tES) treatment that has improved learning and performance in young adults up to nearly 4 times when compared with a sham control. This randomized pilot trial will determine if this same tES protocol improves memory in older adults (50-90 years old) who are healthy, and separately in older adults with mild cognitive impairment (MCI) or early stage Alzheimer's disease (AD). TES will be applied to the right temple and left arm for up to 40 minutes. MRI images, along with other measures, may be obtained before and after tES. If effective, this intervention may help to improve the quality of life for AD patients and their families.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy participants:

1. 50-90 years of age, as verified via photo identification with date of birth.
2. Should be right-handed and learned English by seven years old.
3. Generally healthy

Inclusion criteria for participants with MCI or AD:

1. 50-90 years of age, as verified via photo identification with date of birth.
2. Should be right-handed and learned English by seven years old.
3. Is legally able to sign the consent form on their own behalf, or has a legally authorized representative that is able to sign.
4. Has a caregiver that can assist with taking health history.

Exclusion Criteria:

Exclusion criteria for healthy participants:

1. Significant history of psychiatric disorders or current psychosis including self-report or Geriatric Depression Scale short form score-GDS >5 if uncertain.
2. Current excessive drug, alcohol or nicotine use defined by participant self-report.
3. History of epilepsy, migraines, severe stroke, or traumatic brain injury.
4. Taking medications with significant psychotropic effects.
5. Severe sensory impairment.
6. Severe chronic illness where participation in the study could put participants at an unusual level of risk. Chronic conditions will be evaluated on a case by case basis as they arise.
7. Severe subjective cognitive concerns.
8. Requires a helper animal.
9. Has sufficient prior experience with neurostimulation that might unblind or alter the results.
10. Has metal or electronic implants that may be sensitive to stimulation or could interfere with stimulation or be an MRI contraindication, or has any other MRI contraindication.
11. Has sensitivity to components of tES electrodes being used (typically nickel or latex).
12. Feels ill or have any potential COVID-19 symptoms, such as fever or chills, cough, difficulty breathing, overly tired, unusual aches or pains including headache or sore throat, recent or unusual (for them) loss of taste or smell, congestion or runny nose, nausea or diarrhea.

Exclusion criteria for participants with MCI or AD:

1. Significant history of psychiatric disorders or current psychosis not related to a neurodegenerative condition.
2. Current excessive drug, alcohol or nicotine use.
3. Significant history of epilepsy, stroke, or traumatic brain injury.
4. Taking medications with significant psychotropic effects, not related to neurodegenerative condition
5. Severe sensory impairment
6. Severe chronic illness where participation in the study could put participants at an unusual level of risk. Chronic conditions will be evaluated on a case by case basis as they arise.
7. Requires a helper animal.
8. Has sufficient prior experience with neurostimulation that might unblind or alter the results.
9. Has metal or electronic implants that may be sensitive to stimulation or could interfere with stimulation.
10. Has sensitivity to components of tES electrodes being used (typically nickel or latex).
11. Feels ill or have any potential COVID-19 symptoms, such as fever or chills, cough, difficulty breathing, overly tired, unusual aches or pains including headache or sore throat, unusual loss of taste or smell, or unusual (for them) congestion or runny nose, nausea or diarrhea.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Learning Task Performance | Within one hour after treatment
  Performance accuracy on a complex visual learning and categorization task after full-current tES in comparison to partial-current tES.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Clark, PhD, Principal Investigator — University of New Mexico
Locations (1):
- Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No